CLINICAL TRIAL: NCT06998979
Title: Efficacy of Artificial Intelligence-Generated Music Therapy in Reducing Dental Anxiety Among Adults Undergoing Impacted Third Molar Extraction: A Randomized Controlled Clinical Trial
Brief Title: Efficacy of Artificial Intelligence-Generated Music Therapy in Reducing Dental Anxiety Among Adults Undergoing Impacted Third Molar Extraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Collaborators: University of Salamanca (Other)
Responsible Party: Principal Investigator, Bruno Macedo de Sousa, Professor, University of Coimbra
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: USUCMUSIC2025
Record Dates: First submitted 2025-05-14; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Tooth Extraction; Molar, Third
Keywords: Third molar extraction; Music therapy; Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music therapy (Active Comparator): Patients in the experimental group listened to the music via ambient diffusion from a computer located in the surgical room throughout the entire procedure.
  Interventions: Behavioral: Music therapy
- Control (No Intervention): In the control group, third molar extraction was performed without the application of any music.

INTERVENTIONS:
Behavioral: Music therapy — The music was generated using a beta version of the RIFFUSION program, which is still in its development phase and being refined based on user input. This software operates using neural networks similar to Generative Adversarial Networks (GANs), known as diffusion models. These models begin with random noise and gradually transform it into a musical composition through a process that involves two phases: a diffusion phase-where an existing musical sample is "disordered" by adding random noise-and a reverse phase, in which the noise is removed to reconstruct a new and distinct musical piece.
  The prompt entered into the program was: "Relaxing slow music for people with great stress and extreme anxiety and panic caused by dental surgery with effects of wind and waterfall." A total of 20 songs were generated and merged to achieve a combined duration of 49.20 minutes.
  Arms: Music therapy

SUMMARY:
Music therapy is widely used in dentistry as it helps patients remain distracted during procedures, particularly during implant placement or third molar extraction. This therapy refers to the evidence-based clinical use of music to achieve therapeutic goals, administered by a licensed practitioner. Due to the high prevalence of complications associated with the eruption and development of wisdom teeth, there has been an increase in the rate of surgical extractions, which in turn elevates patients' dental anxiety. Music therapy may aid in the management of anxiety and thereby contribute to a reduction in pain perception. It is a favorable technique due to its low cost and minimal associated risks. In this context, and considering the widespread use of music as a therapeutic tool alongside the emergence of novel technologies-particularly Artificial Intelligence (AI)-this study aims to evaluate the efficacy of AI-generated music therapy in reducing dental anxiety during impacted third molar extraction procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age who provided informed consent
* Patients without severe or uncontrolled systemic diseases
* Patients capable of completing the dental anxiety questionnaires

Exclusion Criteria:

* Patients under 18 years of age
* Patients with severe or uncontrolled systemic diseases
* Patients using anxiolytic medications
* Patients unable to complete the dental anxiety questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-12-04 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Corah's Dental Anxiety Scale | Baseline and immediately after surgery
  The Corah's Dental Anxiety Scale (CDAS) is a reliable instrument for assessing dental anxiety in adults. It consists of four questions addressing different dental situations. Each question is scored on a scale from 1 (not anxious) to 5 (extremely anxious), resulting in a total score ranging from 4 to 20. A score of 15 or higher indicates severe dental anxiety.
Modified Dental Anxiety Scale | Baseline and immediately after surgery
  The Modified Dental Anxiety Scale (MDAS) is a concise, self-administered questionnaire designed to assess levels of dental anxiety. It comprises five items, each rated on a five-point Likert scale ranging from "not anxious" to "extremely anxious." The total score is obtained by summing the individual item scores, yielding a range from 5 to 25.
Spielberger State-Trait Anxiety Inventory | Baseline and immediately after surgery
  The Spielberger State-Trait Anxiety Inventory is a widely recognized psychological instrument for assessing anxiety. It comprises 40 items divided into two subscales: state anxiety, which captures how an individual feels at a particular moment, and trait anxiety, which reflects general, long-term tendencies toward anxiety. Each item is rated on a four-point scale, with higher scores indicating greater levels of anxiety.
Pain Intensity | Immediately after surgery
  To assess perceived pain during the procedure, the Visual Analog Scale (VAS) was used. This scale provides a subjective measure of pain intensity, ranging from 0 to 10, with higher values indicating greater pain.

SECONDARY OUTCOMES:
Body temperature | Baseline and immediately after surgery
  Body temperature reflects the body's ability to regulate heat and maintain homeostasis. It will be measured using a digital thermometer placed axillary (underarm), The body temperature will be measurement in degrees Celsius (°C).
Heart rate | Baseline and immediately after surgery
  Heart rate refers to the number of heartbeats per minute and serves as an indicator of cardiovascular function. It will be measured using a heart rate monitor. The unit of measurement is beats per minute (bpm).
Blood pressure | Baseline and immediately after the surgery
  Blood pressure indicates the force exerted by circulating blood on the walls of the arteries. It will be measured using a digital sphygmomanometer placed around the upper arm. The unit of measurement is millimeters of mercury (mmHg), and it will be recorded as systolic over diastolic pressure (e.g., 120/80 mmHg).
Oxygen saturation | Baseline and immediately after the surgery
  Oxygen saturation refers to the percentage of oxygen-saturated hemoglobin in the blood. It will be measured non-invasively using a pulse oximeter placed on the fingertip. The unit of measurement is percentage (%).

CONTACTS AND LOCATIONS:
Overall Officials: Jose Antonio B Rueda, PhD, Principal Investigator — University of Salamanca
Locations (1):
- Department of Maxillofacial Surgery at the University Hospital Complex of Salamanca, Salamanca, Salamanca, Spain